CLINICAL TRIAL: NCT07131228
Title: Changes in Portal Vein Pulsatility Variability During a Tidal Volume Challenge Can Predict Fluid Tolerance
Acronym: SERLU
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Lucia Valencia, Intensive Care Unit Attending Physician, Dr. Negrin University Hospital
Other Study IDs: DrNegrinUH0000
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Venous Congestion
Keywords: Fluid Responsiveness Fluid Tolerance
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In critically ill patients, appropriate fluid administration is one of the cornerstones of hemodynamic management, as both hypovolemia and fluid overload can negatively impact clinical outcomes.

For years, fluid responsiveness-defined as an increase in cardiac output following volume administration-has guided decision-making in the postoperative ICU. However, fluid responsiveness alone does not guarantee fluid tolerance, which refers to the venous system's ability to accommodate volume without developing venous congestion or adverse effects such as pulmonary edema, renal or hepatic dysfunction.

The tidal volume challenge (TVC)-which consists of a transient increase in tidal volume from 6 to 8 mL/kg-has been shown to predict fluid responsiveness by enhancing the hemodynamic interaction between the heart and lungs during the cardiac cycle, as measured through dynamic arterial indices such as pulse pressure variation (PPV) or stroke volume variation (SVV). However, these indices do not provide information about fluid tolerance or the state of venous congestion.

Doppler ultrasound of the portal vein, specifically the portal pulsatility index (which under normal conditions presents as a continuous waveform due to the damping effects of the hepatic parenchyma and venous compliance), has been proposed as a non-invasive marker of systemic venous congestion. Studies have shown that an increase in the portal pulsatility index following volume loading may indicate the development of venous congestion and, therefore, poor fluid tolerance.

Since the tidal volume challenge transiently increases intrathoracic pressure and allows dynamic evaluation of cardiovascular responses, we propose that this interaction be assessed not only through arterial dynamic indices (which assess responsiveness) but also through changes in venous flow patterns-specifically, variations in portal pulsatility-so that both fluid responsiveness and tolerance can be predicted with the same test.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following:

Age ≥ 18 years at the time of enrollment.

Receiving controlled mechanical ventilation with a baseline tidal volume of 6 mL/kg of predicted body weight.

Clinical indication for assessment of fluid responsiveness.

Adequate acoustic window for ultrasound visualization of the portal vein.

Exclusion Criteria:

Participants will be excluded if they have any of the following:

Liver cirrhosis.

Right heart failure, defined as any of the following on prior echocardiography:

Tricuspid annular plane systolic excursion (TAPSE) < 16 mm

S' wave < 10 cm/s

Right ventricular fractional area change < 35%

Left heart failure (left ventricular ejection fraction < 50%).

Intra-abdominal hypertension.

Atrial fibrillation or other significant cardiac arrhythmias.

Tricuspid regurgitation.

Poor echogenic window preventing adequate ultrasound assessment.

Presence of spontaneous breathing activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective study involving patients admitted to the intensive care unit (ICU) of a tertiary care hospital, who are under mechanical ventilation and present clinical indications for a fluid responsiveness test, such as oliguria or arterial hypotension
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The absolute change in the portal pulsatility index measured in critically ill patients immediately before and after an incraese of voclumen tidal (6 to 8 ml/kg) . Measurements will be obtained using Doppler ultrasonography in vena porta. | Measured immediately before and after the tidal volume challenge (1 minute).

SECONDARY OUTCOMES:
To correlate changes in portal pulsatility during the test with clinical signs of fluid intolerance (e.g., acute kidney injury, pulmonary congestion). | Assessed during the first 48 hours post-challenge.
  The relationship between the change in portal pulsatility index (PPI) during the tidal volume challenge and the occurrence of clinical signs of fluid intolerance in critically ill patients. Clinical signs include acute kidney injury (as defined by KDIGO criteria), pulmonary congestion r lung ultrasound), and other hemodynamic indicators of poor fluid tolerance (proBNP).

IPD SHARING:
Plan to Share IPD: No